CLINICAL TRIAL: NCT04736849
Title: Pilot Study of Epidural and Dorsal Root Stimulation in Humans With Spinal Cord Injury
Brief Title: Epidural and Dorsal Root Stimulation in Humans With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter J. Grahn, Ph.D. (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Peter J. Grahn, Ph.D., Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-006104; 1R01NS115877-01 (NIH)
Record Dates: First submitted 2020-12-18; First posted 2021-02-03 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injuries; Paraplegia; Tetraplegia; Paralysis
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia; Quadriplegia; Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Percutaneous ES and DRS (Experimental): Epidural Stimulation (ES) and Dorsal Root Stimulation (DRS) will be delivered via percutaneously implanted electrodes during rehabilitation. All implanted electrodes will be removed at the end of trial participation. The effects of ES and DRS will be recorded via electrophysiological and biomechanical metrics described within the outcomes measures.
  Interventions: Device: Percutaneous epidural and dorsal root stimulation

INTERVENTIONS:
Device: Percutaneous epidural and dorsal root stimulation — Abbott percutaneous trial lead for dorsal root ganglion neurostimulation (Model MN10350)
  Abbott percutaneous trial lead for epidural neurostimulation (Model 3086)
  Abbott clinician programmer for epidural and dorsal root ganglion neurostimulation (Model 3874)
  Ripple Neuromed Nomad Neurostimulation System

SUMMARY:
A study to compare electrophysiologic activity of epidural stimulation and dorsal root ganglion stimulation, as well as quantify changes in motor performance with both types of stimulation over the course of 10 rehabilitation sessions.

DETAILED DESCRIPTION:
This study aims to expand the understanding of how electrical spinal stimulation enables function, specifically the pathophysiological mechanisms of action underlying spinal electrical stimulation after SCI, and to address the gap in knowledge of spinal sensorimotor network inputs and outputs generated by spinal electrical stimulation in humans with SCI.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury due to trauma located at or above the tenth thoracic vertebrae
* American Spinal Injury Association grading scale of A, B, C, or D
* Intact spinal reflexes below the level of SCI
* SCI must have occurred at least 1 year prior to study enrollment
* At least 22 years of age
* If female, must be willing to use medically-acceptable method of contraception during study participation

Exclusion Criteria:

* Currently a prison inmate, or awaiting trial, related to criminal activity
* Pregnancy at the time of screening for trial enrollment
* Active, untreated urinary tract infection
* Unhealed decubitus ulcer
* Unhealed skeletal fracture
* Spinal abnormality that may impede percutaneous implantation of spinal electrodes
* Untreated clinical diagnosis of psychiatric disorder
* Joint contractures that impede typical range of motion
* Non-MRI-compatible implanted medical devices
* Other implanted stimulation devices (e.g. deep brain stimulator, cardiac pacemaker, diaphragmatic pacer, etc.)
* Undergoing, or planning to undergo, diathermy treatment
* Active participation in an interventional clinical trial
* History of clinically-diagnosed cardiopulmonary disorder, such as severe orthostatic hypotension, which may impede participation in rehabilitation activities such as changes in body position such as supine-to-sit-to-stand activities, prolonged standing, or stepping
* History of frequent and/or severe autonomic dysreflexia
* History of seizure disorder
* Any illness or condition which, based on the research team's assessment, will compromise with the patient's ability to comply with the protocol, patient safety, or the validity of the data collected during this study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Kinematics | Rehabilitation Day 1, Rehabilitation Day 10
  Change in measurements of joint angles, measured in degrees.
Electromyography | Rehabilitation Day 1, Rehabilitation Day 10
  Change in voltage measurements in major muscle groups below the level of injury.
Electroneurography | Rehabilitation Day 1, Rehabilitation Day 10
  Change in voltage measurements from passive electrodes in the epidural space of the lumbar spine and dorsal root nerves.
Foot pressure | Rehabilitation Day 1, Rehabilitation Day 10
  Change in measurements of foot pressure in kilograms through shoe-insole pressure sensors.
Seated pressure | Through study completion, an average of 4 weeks
  Change in measurements of foot pressure in kilograms through a force-sensing array placed beneath the buttocks.
Somatosensory evoked potentials | Through study completion, an average of 4 weeks
  Measurements of change in voltage in the conduction of electricity through the peripheral nerves, cervical and lumbosacral spinal cord, deep brain structures, and sensory cortex, using surface electrodes.
Transcranial magnetic stimulation motor evoked potentials | Through study completion, an average of 4 weeks
  Measurement of change in voltage required to elicit muscle responses in muscle groups known to elicit optimal motor evoked potential responses, both above and below the level of injury.
Injury severity: American Spinal Injury Association Impairment Scale (AIS) | Through study completion, an average of 4 weeks
  Change in measurements of impairment of sensory and motor functions using the American Spinal Injury Association Impairment Scale (AISA Scale). Individuals are classified from A" (complete spinal cord injury) to "E" (normal function). 28 dermatomes and 10 key muscles are assessed bilaterally. Results are summed to produce overall sensory and motor scores and are used in combination with evaluation of anal sensory and motor function as a basis for the determination of AIS classification. Sensory scores are rated 0 (sensation absent) to 2 (normal), bilaterally for each of 28 dermatomes. Muscle function is rated 0 (total paralysis) to 5 (active movement, full range of motion against significant resistance) for each myotome. Upper Extremity Motor Subscores and Lower Extremity Motor Subscores are each scored from 0 to 50; the ASIA Motor Score is scored from 0 to 100. The presence of anal sensation and voluntary anal contraction are assessed as a yes/no.
Patient-reported bowel function | Through study completion, an average of 4 weeks
  Measurement of change in bowel function using the Neurogenic Bowel Dysfunction Score. Answers to qualitative questions are rated from 0 to 5, with a higher number indicating more problematic symptoms, and totaled for a score which categorizes severity of neurogenic bowel symptoms.
Patient-reported bladder function | Through study completion, an average of 4 weeks
  Measurement of change in bladder function using the Neurogenic Bladder Symptom Score. Answers to qualitative questions are rated from 0 to 5, with a higher number indicating more problematic symptoms, and totaled for a score which categorizes severity of neurogenic bladder symptoms.
Male patient-reported sexual function (1) | Through study completion, an average of 4 weeks
  Measurement of change in erectile dysfunction using the Sexual Health Inventory for Men (SHIM). Answers to qualitative questions are rated from 0 to 5, with a higher number indicating better erectile function, and totaled for a score which categorizes severity of erectile dysfunction.
Male patient-reported sexual function (2) | Through study completion, an average of 4 weeks
  Measurement of change in erectile dysfunction using the International Index for Erectile Function (IIEF). Answers to qualitative questions are rated from 0 to 5, with a higher number indicating better erectile function, and totaled for a score which categorizes severity of erectile dysfunction.
Female patient-reported sexual function | Through study completion, an average of 4 weeks
  Measurement of change in sexual function using the Female Sexual Function Index (FSFI). Answers to qualitative questions are rated from 0 to 5, with a higher number indicating better sexual function, and totaled for a score which categorizes severity of sexual dysfunction.
Spasticity | Through study completion, an average of 4 weeks
  Change in measurements of spasticity using the Spinal Cord Injury Spasticity Evaluation Tool (SCI-SET). Answers to qualitative questions are rated from -3 to +3, with a higher positive number indicating more helpful symptoms, and a lower negative number indicating more problematic symptoms. Scores are totaled for a score which categorizes the overall positive or negative impact of a subject's spasticity symptoms.
Neurostimulation user experience | At study completion, an average of 4 weeks
  Rating of the subject's perception of individual aspects of spinal stimulation using the User Experience Questionnaire (UEQ), a survey including 26 descriptive terms and their antonyms. A scoring scale ranging from 1 to 7 determines how closely the subject feels the term or its antonym applies to the intervention, with lower numbers indicating agreement with the term, and higher numbers indicating agreement with the antonym.
Overground ambulation [as appropriate to the subject] (1) | Through study completion, an average of 4 weeks
  Measurement of changes in severity of walking impairment as measured by the Walking Index for Spinal Cord Injury (WISCI II). Trainers combine the type of assistive device(s) used, use or no use of orthotic braces, number of persons assisting ambulation, and distance subject is able to walk (up to 10 meters), into a single score ranging from 0 to 20, with a lower number indicating more severe impairment.
Overground ambulation [as appropriate to the subject] (2) | Through study completion, an average of 4 weeks
  Measurement of changes in overground mobility as measured by the Modified 6 Minute Walk Test. Trainers will assess the distance in meters which the subject can cover in 6 minutes, with a greater distance characterizing better overground mobility.
Balance [as appropriate to the subject] (2) | Through study completion, an average of 4 weeks
  Measurement of changes in ability to perform 14 activities of daily life requiring balance using the Berg Balance Scale. Trainers will assess capabilities in all categories on a 0 to 4 scale, with a higher number indicating greater capability, and total the scores, with a higher total score indicating greater overall balance.
Balance (1) | Through study completion, an average of 4 weeks
  Measurement of changes in basic trunk stability using the Modified Functional Reach Test. Trainers will measure the distance in centimeters the subject can reach forward unsupported without losing trunk stability, with a greater distance indicating greater trunk stability.
Exertion | Through study completion, an average of 4 weeks
  Measurement of change in the subject's psychophysiological exertion using the Borg Rating of Perceived Exertion. Subjects rate the amount of exertion they are experiencing on a rating scale of 6 to 20, with a higher number indicating more exertion.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Grahn, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic-Clinical Trials — https://clinicaltrials.gov/study/NCT04736849

DOCUMENTS (1):
  • Informed Consent Form (2024-08-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT04736849/ICF_000.pdf